CLINICAL TRIAL: NCT00110422
Title: Irbesartan in the Treatment of Hypertensive Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV131-186
Record Dates: First submitted 2005-05-09; First posted 2005-05-10 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2010-06

CONDITIONS: Metabolic Syndrome; Hypertension
Keywords: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Hypertension | interventions — Irbesartan; Hydrochlorothiazide

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: Irbesartan
- B1 (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Irbesartan — Tablets, Oral, 150 mg. titrated to 300 mg, once daily, 28 weeks.
  Other Names: Avapro
  Arms: A1
Drug: Hydrochlorothiazide — Tablets, Oral, 12.5 mg. titrated to 25 mg, once daily, 28 weeks.
  Arms: B1

SUMMARY:
The purpose of this clinical research study is to learn if irbesartan is superior to hydrochlorothiazide relative to effects on insulin sensitivity and glucose metabolism in hypertensive patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to provide written informed consent. Subjects must read, sign, and receive a copy of the informed consent prior to any study procedures, including withdrawal of any antihypertensive medication.
* Males and females >= 18 years of age.
* Uncontrolled hypertension defined as an average systolic blood pressure >= 140 mmHg and/or an average diastolic blood pressure >= 90 mmHg. This applies to both people not taking any blood pressure medications and people taking just one blood pressure medication.
* Presenting at least 2 of the following:

  * Obesity;
  * High triglycerides;
  * Low HDL cholesterol;
  * Elevated fasting glucose.

Exclusion Criteria:

* Women of child bearing potential who are not using adequate birth control.
* Women who are pregnant or breastfeeding
* Diabetics
* Systolic blood pressure >= 180 mmHg.
* Diastolic blood pressure >= 110 mmHg.
* Stroke within past 12 months.
* Myocardial infarction and heart revascularization procedure or acute angina within past 6 months.
* Moderate to severe heart failure.
* Significant kidney or liver disease.
* Cancer in past 5 years.
* Drug or alcohol abuse.
* Gout
* Lupus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin resistance(MatsudaIndex)Week16

SECONDARY OUTCOMES:
Change from baseline in insulin resist-QuickiIndex Week16;Change from baseline in triglyc.,BP,hs-CRP,albumin/creatinine ratio Week16;Changes from baseline-Matsuda,QuickiIndex,BP,triglyc.,hs-CRP&albumin/creatinine ratio Week28

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- France (3):
  - Local Institution, Angers
  - Local Institution, Nantes
  - Local Institution, Tiercé
- Germany (6):
  - Local Institution, Hanover
  - Local Institution, München
  - Local Institution, Ornbau
  - Local Institution, Rotenburg An de Fluda
  - Local Institution, Tübingen
  - Local Institution, Villingen-Schwenningen
- Italy (5):
  - Local Institution, Ancona
  - Local Institution, Chieti Scalo
  - Local Institution, Pisa
  - Local Institution, Ravenna
  - Local Institution, Sassari
- Norway (2):
  - Local Institution, Oslo
  - Local Institution, Snaroya
- Russia (4):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Yaroslavl
- Spain (5):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Granada
  - Local Institution, Seville
  - Local Institution, Zaragoza

REFERENCES:
- [Background] Parhofer KG, Birkeland KI, DeFronzo R, Del Prato S, Bhaumik A, Ptaszynska A. Irbesartan has no short-term effect on insulin resistance in hypertensive patients with additional cardiometabolic risk factors (i-RESPOND). Int J Clin Pract. 2010 Jan;64(2):160-8. doi: 10.1111/j.1742-1241.2009.02246.x. Epub 2009 Nov 19. PMID 19929980